CLINICAL TRIAL: NCT06706817
Title: A Multicentre, Single-Arm, Phase 3b Study to Assess Changes in Symptoms in Adult Participants With Chronic Rhinosinusitis With Nasal Polyposis Initiating Treatment With Tezepelumab (ESSENCE)
Brief Title: A Study to Investigate Changes in Symptoms in Adult Participants With Chronic Rhinosinusitis With Nasal Polyposis Initiating Treatment With Tezepelumab
Acronym: ESSENCE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Fortrea (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5242C00002
Record Dates: First submitted 2024-11-07; First posted 2024-11-27 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps
Keywords: Chronic rhinosinusitis; Rhinosinusitis
MeSH Terms: conditions — Rhinosinusitis | interventions — tezepelumab

STUDY DESIGN:
Intervention Model Description: Open-Label, single-arm treatment study. Participants will be treated with tezepelumab Q4W from Week 0, with the last dose administered at Week 20
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Tezepelumab (Experimental): Tezepelumab: Tezepelumab single dose subcutaneously injection.
  Interventions: Combination Product: Tezepelumab

INTERVENTIONS:
Combination Product: Tezepelumab — IMP. Subcutaneous injection. Unit dose strengths 210 mg.
  Other Names: TEZSPIRE®

SUMMARY:
The main objective of this study is to evaluate treatment outcomes of tezepelumab among participants with physician-determined surgery-eligible CRSwNP, with or without asthma.

Study details include:

1. The study duration will be up to 40 weeks.
2. The treatment duration will be up to 24 weeks.
3. The visit frequency will be once every 4 weeks (Q4W).

DETAILED DESCRIPTION:
This is a multicentre, open-label, single-arm, phase IIIb study is to describe changes from baseline in (1) participant-reported nasal congestion as evaluated by the nasal congestion score (NCS) and (2) participant-reported sino-nasal symptoms as evaluated by sino-nasal outcome test, 22 item (SNOT-22) following initiation of tezepelumab treatment.

Approximately 60 sites in 10 countries will enrol adult patients with physician determined surgery eligible CRSwNP.

The study is divided into 3 periods as described below:

* Screening Period (from Week -4 until Week 0, up to 4 Weeks)
* Treatment period (Week 0 to Week 24)
* Safety Follow-up Period (Week 24 to Week 36)

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years of age or older, at the time of signing the informed consent.
* Participants with physician-diagnosed CRSwNP for at least 12 months prior to Visit 1 who have all of the following:
* Severity consistent with the need for surgery as defined by total NPS ≥ 4 (at least 2 for each nostril) at screening, as determined by the central reader
* Mean NCS ≥ 2 in the 2 weeks prior to Visit 2
* Ongoing documented NP symptoms for > 8 weeks prior to screening such as rhinorrhoea, reduction or loss of smell and/or poor quality/loss of sleep
* SNOT-22 total score ≥ 30 as assessed at screening. Note: approximately 50 participants with a NPS = 4 at screening will receive treatment with tezepelumab.
* Any standard of care for treatment of CRSwNP, which must include treatment with intranasal corticosteroids, provided the participant is stable on that treatment for at least 30 days prior to Visit 1. Investigators should also assure that participants are compliant and on a stable dose of the background INCS during study period.
* Either 1) documented treatment of NP exacerbation with SCS for at least 3 consecutive days or one IM depo-injectable dose (or contraindications/intolerance to) within the past 12 months prior to Visit 1 but not within the last 3 months prior to Visit 1 OR 2) any history of NP surgery (or contraindications/intolerance to)
* Body weight of ≥ 40 kg at Visit 1
* Female participants:
* Contraceptive use by women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. Women of non childbearing potential are defined as women who are either permanently sterilised (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy), or who are postmenopausal.
* Women will be considered postmenopausal if they have been amenorrhoeic for 12 months prior to the planned start date of the first IMP administration without an alternative medical cause.

The following age-specific requirements apply:

* Women < 50 years old would be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatment and FSH levels in the postmenopausal range.
* Women ≥ 50 years old would be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of all exogenous hormonal treatment.
* WOCBP must be willing to use one of the methods of contraception described hereafter, from the time of signing the ICF throughout the study and 16 weeks after last tezepelumab administration:
* Combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal, transdermal
* Progestogen-only hormonal contraception associated with inhibition of ovulation: oral, injectable, implantable
* Intrauterine device
* Intrauterine hormone-releasing system
* Bilateral tubal occlusion
* Vasectomised partner (vasectomised partner is a highly effective birth control method provided that the partner is the sole sexual partner of the WOCBP participant and that the vasectomised partner has received medical assessment of the surgical success)
* Sexual abstinence: it is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the participant.
* Cessation of contraception after this point should be discussed with a responsible physician.
* Provision of signed and dated written ICF as described in Appendix A 3 prior to any mandatory study-specific procedures, sampling, and analyses.
* Participant who is capable of giving signed informed consent as described in Appendix A 3 which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

Exclusion Criteria:

* Participants with documented allergic fungal rhinosinusitis and/or central compartment atopic disease.
* Any clinically important pulmonary disease other than asthma (eg, active lung infection, bronchiectasis, pulmonary fibrosis, cystic fibrosis, primary ciliary dyskinesia, allergic bronchopulmonary mycosis, hypereosinophilic syndromes, etc) that could confound interpretation of clinical CRSwNP endpoints results.
* Any disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, haematological, psychiatric, or major physical impairment that is not stable in the opinion of the investigator and could:

  * Affect the safety of the participant throughout the study
  * Influence the findings of the study or the interpretation
  * Impede the participant's ability to complete the entire duration of study.
* Sinus surgery within 6 months of screening visit OR any sinus surgery in the past which changed the lateral wall of the nose making NPS evaluation impossible.
* Participants with conditions or concomitant disease that makes them non-evaluable for the primary CRSwNP endpoints such as:
* Antrochoanal polyps
* Nasal septal deviation that occludes at least one nostril
* Acute sinusitis, nasal infection, asthma exacerbation or upper respiratory infection at screening or in the two weeks before screening, or Churg-Strauss syndrome (also known as eosinophilic granulomatosis with polyangiitis), Young's syndrome or Kartagener's syndrome
* History of cancer:

  1. Participants who have had basal cell carcinoma, localised squamous cell carcinoma of the skin or in situ carcinoma of the cervix are eligible to participate in the study provided that curative therapy was completed at least 12 months prior to Visit 1.
  2. Participants who have had other malignancies are eligible provided that curative therapy was completed at least 5 years prior to Visit 1.
* Uncontrolled epistaxis within 2 months of Visit 1
* A helminth parasitic infection diagnosed within 6 months prior to Visit 1 that has not been treated with, or has failed to respond to, standard of care therapy.
* For participants with comorbid asthma: Current smokers or participants with a smoking history ≥ 10 packs per year and participants using vaping products, including electronic cigarettes. Former smokers with a smoking history of < 10 pack per year and users of vaping or e-cigarette products must have stopped for at least 6 months prior to Visit 1 to be eligible.
* History of chronic alcohol or drug abuse within 12 months prior to Visit 1.
* Tuberculosis requiring treatment within the 12 months prior to Visit 1.
* Major surgery within 8 weeks prior to Visit 1 or planned NP surgery or planned surgical procedures requiring general anaesthesia or inpatient status for more than 1 day during the conduct of the study.
* History of known immunodeficiency disorder including a positive HIV test at Visit 1, or the participant taking antiretroviral medications as determined by medical history and/or participant's verbal report.
* Infection requiring systemic antibiotics within 14 days prior to Visit 1. Note: Participants with respiratory infections requiring antibiotics within 14 days prior to Visit 1 may extend their screening period to allow recovery and return no sooner than 14 days after completion of therapy.
* Evidence of COVID-19 within 4 weeks prior to screening or ongoing clinically significant COVID-19 sequelae (eg, participants who have long-term post-COVID-19 anosmia).
* Receipt of any marketed or investigational biologic agent within 4 months or 5 half-lives (whichever is longer) prior to Visit 1 or receipt of any investigational non-biologic agent within 30 days or 5 half-lives (whichever is longest) prior to Visit 1.
* Treatment with systemic immunosuppressive/immunomodulating drugs (eg, methotrexate, cyclosporine, etc.), except for SCS used in the treatment of asthma/asthma exacerbations, within the last 12 weeks or 5 half-lives (whichever is longer) prior to Visit 1.
* Receipt of immunoglobulin or blood products within 30 days prior to Visit 1.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2027-01-29 (Estimated); Study Completion 2027-01-29 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in nasal congestion | Week 24
  Changes from baseline in participant-reported nasal congestion as evaluated by the nasal congestion score (NCS) as part of the nasal polyposis symptom diary (NPSD) following initiation of tezepelumab treatment.
Change from baseline in sino-nasal symptoms | Week 24
  changes from baseline in participant reported sino nasal symptoms as evaluated by sino nasal outcome test, 22 item (SNOT 22) total score following initiation of tezepelumab treatment.

SECONDARY OUTCOMES:
Proportion of NCS responders | End of treatment - Week 24
  Proportion of NCS responders (minimal clinically important difference [MCID] from baseline = 1.0) at each collected timepoint.
Time to first response for NCS | End of Treatment-week 24
  Description of time to first response for NCS by analysing data at all collected timepoints.
Change from baseline in NCS | Daily for the 2 weeks prior to Week 0 through end of treatment visit (EOT; Week 24).
  Change from baseline in NCS at each collected timepoint.
Proportion of SNOT-22 responders | Screening, Weeks 0, 2, 4, 8, 12, 16, 20, and 24.
  Proportion of SNOT-22 responders (MCID from baseline = -8.9) at each collected timepoint.
Time to first response for SNOT-22 | Screening, Weeks 0, 2, 4, 8, 12, 16, 20, and 24.
  Description of time to first response for SNOT-22 by analysing data at all collected timepoints.
Change from baseline in SNOT-22 | Screening, Weeks 0, 2, 4, 8, 12, 16, 20, and 24.
  Change from baseline in SNOT-22 at each collected timepoint.
Change from baseline visit in nasal blockage (NB) | Weeks 0, 4, 12, and 24.
  Change from baseline visit in NB measured by PNIF
Change from baseline visit in NB | daily for the 2 weeks prior to Week 0 through the first 12 weeks of Treatment Period, and at Weeks 16, 20, 24.
  Change from baseline visit in NB measured by VAS-NB
Proportion of PNIF responders | Weeks 0, 4, 12, and 24.
  Proportion of PNIF responders (MCID from baseline =20 L/min).
Proportion of VAS-NB responders | daily for the 2 weeks prior to Week 0 through the first 12 weeks of Treatment Period, and at Weeks 16, 20, 24.
  Proportion of VAS-NB responders (MCID from baseline = -3.0) (in participants with VAS-NB ≥ 7 at baseline).
Time to first response for PNIF | Weeks 0, 4, 12, and 24
  Description of time to first response for PNIF by analysing data at all collected timepoints.
First response for VAS NB | daily for the 2 weeks prior to Week 0 through the first 12 weeks of Treatment Period, and at Weeks 16, 20, 24.
  Description of time to first response for VAS NB by analysing data at all collected timepoints (in participants with VAS-NB ≥ 7 at baseline).
Change from baseline in loss of smell score evaluated by UPSIT or Sniffin Sticks | Weeks 0, 1, 2, 4, 8, 12, 16, 20, and 24
  Change from baseline in loss of smell score evaluated by UPSIT or Sniffin Sticks
Change from baseline in loss of smell score evaluated by VAS-Taste | daily for the 2 weeks prior to Week 0 through the first 12 weeks of Treatment Period, and at Weeks 16, 20, and 24
  Change from baseline in loss of smell score evaluated by VAS-Taste
Change from baseline in loss of smell score evaluated by VAS-Smell | daily for the 2 weeks prior to Week 0 through the first 12 weeks of Treatment Period, and at Weeks 16, 20, and 24.
  Change from baseline in loss of smell score evaluated by VAS-Smell
Proportion of UPSIT responders | Weeks 0, 1, 2, 4, 8, 12, 16, 20, and 24.
  Proportion of UPSIT responders (MCID from baseline = 4)
Proportion of Sniffin sticks responders | Weeks 0, 1, 2, 4, 8, 12, 16, 20, and 24
  Proportion of Sniffin sticks responders (MCID from baseline = 6)
Proportion of VAS-Smell responders | daily for the 2 weeks prior to Week 0 through the first 12 weeks of Treatment Period, and at Weeks 16, 20, and 24
  Proportion of VAS-Smell responders (MCID from baseline = -3.0) (in participants with VAS-Smell ≥ 7 at baseline)
Proportion of participants with a reduction in VAS-Taste score from baseline | daily for the 2 weeks prior to Week 0 through the first 12 weeks of Treatment Period, and at Weeks 16, 20, and 24.
  Proportion of participants with a reduction in VAS-Taste score from baseline (in participants with VAS-Taste ≥ 7 at baseline)
Time to first response for UPSIT/Sniffin sticks | Weeks 0, 1, 2, 4, 8, 12, 16, 20, and 24
  Time to first response for UPSIT/Sniffin sticks by analysing data at all collected timepoints.
Time to first response for VAS Smell | daily for the 2 weeks prior to Week 0 through the first 12 weeks of Treatment Period, and at Weeks 16, 20, and 24
  Time to first response for VAS Smell by analysing data at all collected timepoints (in participants with VAS-Smell ≥ 7 at baseline).
Time to first improvement in VAS-Taste | daily for the 2 weeks prior to Week 0 through the first 12 weeks of Treatment Period, and at Weeks 16, 20, and 24.
  Time to first improvement in VAS-Taste by analysing data at all collected timepoints (in participants with VAS-Taste ≥ 7 at baseline).
Change from baseline in sleep as evaluated by PSQI total score | Weeks 0, 12, and 24.
  Change from baseline in sleep as evaluated by PSQI total score
Change from baseline in sleep as evaluated by SNOT-22 Sleep domain score | Screening, Week 0, Weeks 2, 4, 8, 12, 16, 20, and 24
  Change from baseline in sleep as evaluated by SNOT-22 Sleep domain score
Change from baseline in sleep as evaluated by VAS-Sleep | daily for the 2 weeks prior to Week 0 through the first 12 weeks of Treatment Period, and at Weeks 16, 20, and 24
  Change from baseline in sleep as evaluated by VAS-Sleep
Proportion of PSQI responders | Weeks 0, 12, and 24
  Proportion of PSQI responders (MCID from baseline = - 4.4)
Proportion of SNOT-22 Sleep domain responders | Screening, Week 0, Weeks 2, 4, 8, 12, 16, 20, and 24
  Proportion of SNOT-22 Sleep domain responders (MCID from baseline = -2.9)
Proportion of participants with any improvement in VAS Sleep from baseline | Daily for the 2 weeks prior to Week 0 through the first 12 weeks of Treatment Period, and at Weeks 16, 20, and 24
  Proportion of participants with any improvement in VAS Sleep from baseline (in participants with VAS-Sleep ≥ 7 at baseline)
Time to first response for PSQI | Weeks 0, 12, and 24.
  Time to first response for PSQI by analysing data at all collected timepoints.
Time to first response for SNOT-22 Sleep domain | Screening, Week 0, Weeks 2, 4, 8, 12, 16, 20, and 24.
  Time to first response for SNOT-22 Sleep domain by analysing data at all collected timepoints.
Time to first improvement for VAS-Sleep | daily for the 2 weeks prior to Week 0 through the first 12 weeks of Treatment Period, and at Weeks 16, 20, and 24
  Time to first improvement for VAS-Sleep by analysing data at all collected timepoints (in participants with VAS-Sleep ≥ 7 at baseline).
Change from baseline in total NPS | Screening, Weeks 2 and 24
  Change from baseline in total NPS evaluated by nasal endoscopy.
Proportion of NPS responders | Screening, Weeks 2 and 24
  Proportion of NPS responders (MCID from baseline = 1.0) at Weeks 2 and 24.
Change from baseline in NPQ score | Weeks 0, 8, 12, and 24.
  Change from baseline in NPQ score
Proportion of NPQ responders | Weeks 0, 8, 12, and 24
  Proportion of NPQ responders (MCID from baseline = 7.0)
Time to first response for NPQ | Weeks 0, 8, 12, and 24.
  Time to first response for NPQ by analysing data collected at each specified timepoint.
Change from baseline in TSS | daily for the 2 weeks prior to Week 0 and through EOT (Week 24)
  Change from baseline in TSS
Proportion of TSS responders | daily for the 2 weeks prior to Week 0 and through EOT (Week 24)
  Proportion of TSS responders (MCID from baseline = 4.0)
Time to first response for TSS | daily for the 2 weeks prior to Week 0 and through EOT (Week 24)
  Time to first response for TSS by analysing data at all collected timepoints.
Change from baseline in NP severity | daily for the 2 weeks prior to Week 0 through the first 12 weeks of Treatment Period, and at Weeks 16, 20, and 24.
  Change from baseline in NP severity as measured by VAS Overall symptoms
Proportion of VAS Overall symptom responders | daily for the 2 weeks prior to Week 0 through the first 12 weeks of Treatment Period, and at Weeks 16, 20, and 24.
  Proportion of VAS Overall symptom responders (MCID from baseline = 2.5)
Time to first response for VAS-Overall symptom | daily for the 2 weeks prior to Week 0 through the first 12 weeks of Treatment Period, and at Weeks 16, 20, and 24.
  Time to first response for VAS-Overall symptom by analysing data at all collected timepoints
Proportion of participants who respond as 'well controlled' or 'completely controlled' NP symptoms to the NP control question | Weeks 0, 4, 8, 12, 20, and 24.
  Proportion of participants who respond as 'well controlled' or 'completely controlled' NP symptoms to the NP control question
Time to first response for NP control | Weeks 0, 4, 8, 12, 20, and 24.
  Time to first response for NP control by analysing data at all collected timepoints.

OTHER OUTCOMES:
Endoscopy findings will be used to describe histological changes and describe CRSwNP visualization | Screening, Weeks 2 and 24
  Endoscopy findings will be used to describe histological changes and describe CRSwNP visualization from baseline to Week 24.
Change from baseline in blood eosinophil count (BEC), total serum IgE, specific IgE (including fungi/moulds [eg, Alternaria]), S. aureus enterotoxin IgE, and Fractional exhaled nitric oxide (FeNO; for asthma participants only) | Screening (for BEC and FeNO), Week 0 (for IgE and S. aureus enterotoxin IgE), Weeks 12 and 24
  Change from baseline in blood eosinophil count (BEC), total serum IgE, specific IgE (including fungi/moulds [eg, Alternaria]), S. aureus enterotoxin IgE, and Fractional exhaled nitric oxide (FeNO; for asthma participants only)
Change from baseline in WPAI-CRSwNP | Week 0 and Week 24
  Change from baseline in WPAI-CRSwNP
Proportion and annualised rate of primary care visits (all rates for CRSwNP-related and asthma-related). | 24 weeks pre-and post index (index = 1st tezepelumab dosing).
  Proportion and annualised rate of primary care visits (all rates for CRSwNP-related and asthma-related).
Change in incident rate of nasal infection comparing the post-index period versus the pre-index period | 24 weeks pre- and post-index. (index = 1st tezepelumab dosing)
  Change in incident rate of nasal infection comparing the post-index period versus the pre-index period (index = 1st tezepelumab dosing).
Change in proportion of participants with CRSwNP-related SCS use during the post-index period (24 weeks following tezepelumab first dose) versus the pre-treatment period (24 weeks prior to tezepelumab first dose) | 24-weeks pre- and post- index. (index = 1st tezepelumab dosing).
  Change in proportion of participants with CRSwNP-related SCS use during the post-index period (24 weeks following tezepelumab first dose) versus the pre-treatment period (24 weeks prior to tezepelumab first dose)
Change in average SCS daily dose during the post-index period versus dose at/closest to the index | 24-weeks pre- and post- index. (index = 1st tezepelumab dosing).
  Change in average SCS daily dose during the post-index period (24 weeks following tezepelumab first dose) versus dose at/closest to the index
Proportion of participants with the decision for CRSwNP surgery during the 24 weeks pre- and post-index and change in NP surgery proportion following tezepelumab initiation. | 24-weeks pre- and post- index. (index = 1st tezepelumab dosing).
  Proportion of participants with the decision for CRSwNP surgery during the 24 weeks pre- and post-index and change in NP surgery proportion following tezepelumab initiation.
Proportion of patients with CRSwNP exacerbation | 24-weeks pre- and post-index (index = 1st tezepelumab dosing).
  Proportion of patients with CRSwNP exacerbation
Change since baseline in Asthma Control Questionnaire 6 (ACQ-6) score | Weeks 0 and 24.
  Change since baseline in Asthma Control Questionnaire 6 (ACQ-6) score
ACQ-6 responder: proportion of participants with change since baseline in ACQ-6 of 0.5 or above | Weeks 0 and 24
  ACQ-6 responder: proportion of participants with change since baseline in ACQ-6 of 0.5 or above
Annualised asthma exacerbation rate | 24 weeks pre-and post-index (index = 1st tezepelumab dosing).
  Annualised asthma exacerbation rate
Change from baseline in Annualised asthma exacerbation rate | 24 weeks pre-and post-index (index = 1st tezepelumab dosing).
  Change from baseline in Annualised asthma exacerbation rate
Lung function (Forced expiratory volume in 1 second [FEV1]) (if available at site) | Weeks 0, 12 (lung function only) and 24.
  Lung function (Forced expiratory volume in 1 second [FEV1]) (if available at site)
Asthma-related SCS use (yes/no) | 24 weeks pre-and post-index (index = 1st tezepelumab dosing).
  Asthma-related SCS use (yes/no)
Proportion and annualised rate of urgent care (all rates for CRSwNP-related and asthma-related). | 24 weeks pre-and post index (index=1st tezepelumab dosing)
  Proportion and annualised rate of urgent care (all rates for CRSwNP-related and asthma-related).
Proportion and annualised rate of unplanned surgery (all rates for CRSwNP-related and asthma-related). | 24 weeks pre and post index (index=ist tezepelumab dosing)
  Proportion and annualised rate of unplanned surgery (all rates for CRSwNP-related and asthma-related).
Proportion and annualised rate of unplanned out participant visits (all rates for CRSwNP-related and asthma-related). | 24 weeks pre- and post index (index=1st tezepelumab dosing)
  Proportion and annualised rate of unplanned out participant visits (all rates for CRSwNP-related and asthma-related).
Proportion and annualised rate of emergency room visits (all rates for CRSwNP-related and asthma-related). | 24 weeks pre-and post index (index=1st tezepelumab dosing)
  Proportion and annualised rate of emergency room visits (all rates for CRSwNP-related and asthma-related).
Proportion and annualised rate of hospitalisations (all rates for CRSwNP-related and asthma-related). | 24 weeks pre-and post index(index=1st tezepelumab dosing)
  Proportion and annualised rate of hospitalisations (all rates for CRSwNP-related and asthma-related).
Asthma related SCS use as part of an exacerbation | 24 weeks pre-and post index(index=1st tezepelumab dosing)
  Asthma related SCS use as part of an exacerbation
Asthma related SCS duration of use | 24 weeks pre-and post index(index=1st tezepelumab dosing)
  Asthma related SCS duration of use
Asthma related SCS daily dose | 24 weeks pre-and post index(index=1st tezepelumab dosing)
  Asthma related SCS daily dose

CONTACTS AND LOCATIONS:
Overall Officials: Tanya M Laidlaw, MD, Principal Investigator — Director of Translational Research in Allergy and Director of the Aspirin-Exacerbated Respiratory Disease (AERD) Centre at the Brigham and Women's Hospital.; Enrico Heffler, MD, PhD, Principal Investigator — Associate Professor of Internal Medicine and Consultant at the Personalized Medicine, Asthma and Allergy Unit at IRCCS Humanitas Research Hospital
Locations (40):
- United States (4):
  - Research Site, Newport Beach, California
  - Research Site, Chicago, Illinois
  - Research Site, Chestnut Hill, Massachusetts
  - Research Site, Columbia, Missouri
- Bulgaria (2):
  - Research Site, Plovdiv
  - Research Site, Sofia
- Canada (2):
  - Research Site, Hamilton, Ontario
  - Research Site, Québec, Quebec
- France (7):
  - Research Site, Le Kremlin-Bicêtre
  - Research Site, Lille
  - Research Site, Marseille
  - Research Site, Nantes
  - Research Site, Pierre-Bénite
  - Research Site, Poitiers
  - Research Site, Toulouse
- Germany (5):
  - Research Site, Düsseldorf
  - Research Site, Marburg
  - Research Site, Tübingen
  - Research Site, Villingen-Schwenningen
  - Research Site, Wiesbaden
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Nyíregyháza
  - Research Site, Pécs
- Italy (8):
  - Research Site, Bologna
  - Research Site, Catania
  - Research Site, Florence
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Rozzano
- Poland (4):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Lodz
  - Research Site, Zawadzkie
- Spain (5):
  - Research Site, Barcelona
  - Research Site, Cadiz
  - Research Site, Madrid
  - Research Site, Salamanca
  - Research Site, Santiago de Compostela

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/